CLINICAL TRIAL: NCT00002533
Title: A PHASE II/III PILOT STUDY OF THE EFFECTS OF PROPHYLACTIC FLUCONAZOLE THERAPY ON MUCOSITIS IN PATIENTS UNDERGOING RADIATION TREATMENT FOR HEAD AND NECK CANCER
Brief Title: Fluconazole in Preventing Mucositis in Patients Undergoing Radiation Therapy for Head and Neck Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 19920577; CDR0000078457 (Registry Identifier: PDQ (Physician Data Query)); NCI-V93-0288; SCCC-1992110 (Other: University of Miami Sylvester Comprehensive Cancer Center)
Record Dates: First submitted 1999-11-01; First posted 2003-09-18 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Head and Neck Cancer; Infection; Oral Complications
Keywords: untreated metastatic squamous neck cancer with occult primary; recurrent metastatic squamous neck cancer with occult primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma; oral complications; stage I squamous cell carcinoma of the lip and oral cavity; stage I basal cell carcinoma of the lip; stage I verrucous carcinoma of the oral cavity; stage I mucoepidermoid carcinoma of the oral cavity; stage I adenoid cystic carcinoma of the oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage II basal cell carcinoma of the lip; stage II verrucous carcinoma of the oral cavity; stage II mucoepidermoid carcinoma of the oral cavity; stage II adenoid cystic carcinoma of the oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage III basal cell carcinoma of the lip; stage III verrucous carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV basal cell carcinoma of the lip; stage IV verrucous carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent verrucous carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; stage I squamous cell carcinoma of the oropharynx; stage I lymphoepithelioma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage II lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent lymphoepithelioma of the oropharynx; stage I squamous cell carcinoma of the nasopharynx; stage I lymphoepithelioma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage II lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the nasopharynx; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the larynx; stage I verrucous carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage I inverted papilloma of the paranasal sinus and nasal cavity; stage I midline lethal granuloma of the paranasal sinus and nasal cavity; stage I esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II inverted papilloma of the paranasal sinus and nasal cavity; stage II midline lethal granuloma of the paranasal sinus and nasal cavity; stage II esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; infection
MeSH Terms: conditions — Head and Neck Neoplasms; Infections; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory | interventions — Fluconazole; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: fluconazole
Radiation: radiation therapy

SUMMARY:
RATIONALE: Giving fluconazole may be effective in preventing or controlling mucositis caused by radiation therapy to the head and neck.

PURPOSE: Randomized phase II/III trial to study the effectiveness of fluconazole in preventing mucositis in patients undergoing radiation therapy for head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the effect of prophylactic antifungal therapy with fluconazole on the incidence and severity of radiation-associated mucositis/thrush in patients with head and neck cancer undergoing definitive radiotherapy.

OUTLINE: This is a randomized study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo standard hyperfractionated radiotherapy 5 days a week for 5-5.6 weeks. Patients receive oral fluconazole on days 1-4 and 28-31 of radiotherapy.
* Arm II: Patients undergo radiotherapy as in arm I. Patients who develop a microbiologically proven fungal infection or clinically evident oral cavity and/or oropharyngeal thrush may receive fluconazole as in arm I.

PROJECTED ACCRUAL: At least 42 patients (26 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven head and neck cancer undergoing definitive radiotherapy

PATIENT CHARACTERISTICS:

Age:

* Over 21

Performance status:

* Karnofsky 70-100%

Hematopoietic:

* Not specified

Hepatic:

* SGOT and SGPT less than 2 times normal
* Alkaline phosphatase less than 2 times normal

Renal:

* Not specified

Other:

* No history of hypersensitivity to fluconazole
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* At least 2 months since prior antifungal agents
* Not currently receiving phenytoin, hydrochlorothiazide, or warfarin

  * If these medications are initiated during study therapy, medication serum levels and electrolytes are monitored for possibility of drug interaction

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1993-02; Primary Completion 2006-06 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnold M. Markoe, MD, ScD, Study Chair — University of Miami Sylvester Comprehensive Cancer Center
Locations (1):
- Sylvester Cancer Center, University of Miami, Miami, Florida, United States